CLINICAL TRIAL: NCT01548144
Title: A Two Steps Phase I Trial of Pazopanib or Pemetrexed in Combination With Crizotinib Followed by the Triplet, Crizotinib Plus Pazopanib Plus Pemetrexed in Patients With Advanced Malignancies
Brief Title: Pazopanib or Pemetrexed and Crizotinib in Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI request
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-1142; NCI-2012-00324 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancers; Advanced Malignancies; Crizotinib; PF-02341066; Pazopanib; Gw786034; Pemetrexed; LY231514; Alimta; MTA; Multitargeted Antifolate; NSC-698037
MeSH Terms: interventions — Crizotinib; pazopanib; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Crizotinib + Pazopanib - Group A (Experimental): Starting dose for Crizotinib: 250 mg by mouth every other day, 1 or 2 times a day on Day 1 of a 21 day cycle. Participant told how often to take this drug.
  Dose Expansion Group: MTD from Phase 1.
  Starting Dose for Pazopanib: 200 mg by mouth daily in a 21 day cycle.
  Dose Expansion Group: MTD from Phase 1.
  Interventions: Drug: Crizotinib (Xalkori); Drug: Pazopanib
- Crizotinib + Pemetrexed - Group B (Experimental): Starting dose for Crizotinib: 250 mg by mouth every other day, 1 or 2 times a day on Day 1 of a 21 day cycle. Participant told how often to take this drug.
  Dose Expansion Group: MTD from Phase 1.
  Starting dose for Pemetrexed: 200 mg/m2 by vein every 3 weeks on Day 1 of a 21 day cycle.
  Dose Expansion Group: MTD from Phase 1.
  Interventions: Drug: Crizotinib (Xalkori); Drug: Pemetrexed
- Pazopanib + Pemetrexed - Group C (Experimental): Starting dose for Pazopanib: 200 mg by mouth daily in a 21 day cycle.
  Expansion group starting dose: MTD from Phase 1.
  Starting dose for Pemetrexed: 200 mg/m2 by vein on Day 1 of a 21 day cycle.
  Expansion group starting dose: MTD from Phase 1.
  Interventions: Drug: Pazopanib; Drug: Pemetrexed
- Crizotinib + Pazopanib + Pemetrexed - Group D (Experimental): Starting dose for Crizotinib: 250 mg by mouth every other day, 1 or 2 times a day on Day 1 of a 21 day cycle. Participant told how often to take this drug.
  Dose Expansion Group: MTD from Phase 1.
  Starting Dose for Pazopanib: 200 mg by mouth daily in a 21 day cycle.
  Dose Expansion Group: MTD from Phase 1.
  Starting dose for Pemetrexed: 400 mg/m2 by vein every 3 weeks on Day 1 of a 21 day cycle.
  Dose Expansion Group: MTD from Phase 1.
  Interventions: Drug: Crizotinib (Xalkori); Drug: Pazopanib; Drug: Pemetrexed

INTERVENTIONS:
Drug: Crizotinib (Xalkori) — Starting dose for Crizotinib - Groups A, B, C: 250 mg by mouth every other day, 1 or 2 times a day on Day 1 of a 21 day cycle. Participant told how often to take this drug.
  Expansion Groups Starting Dose: MTD from Phase 1.
  Other Names: PF-02341066; Xalkori
  Arms: Crizotinib + Pazopanib + Pemetrexed - Group D; Crizotinib + Pazopanib - Group A; Crizotinib + Pemetrexed - Group B
Drug: Pazopanib — Starting Dose for Pazopanib - Groups A, C, D: 200 mg by mouth daily in a 21 day cycle.
  Expansion Groups Starting Dose: MTD from Phase 1.
  Other Names: GW786034
  Arms: Crizotinib + Pazopanib + Pemetrexed - Group D; Crizotinib + Pazopanib - Group A; Pazopanib + Pemetrexed - Group C
Drug: Pemetrexed — Starting dose for Pemetrexed - Groups B + C: 200 mg/m2 by vein on Day 1 of a 21 day cycle.
  Expansion Groups Starting Dose: MTD from Phase 1.
  Starting dose for Pemetrexed Group D: 400 mg/m2 by vein every 3 weeks on Day 1 of a 21 day cycle.
  Expansion Group Starting Dose: MTD from Phase 1.
  Other Names: LY231514; Alimta; MTA; Multitargeted Antifolate; NSC-698037
  Arms: Crizotinib + Pazopanib + Pemetrexed - Group D; Crizotinib + Pemetrexed - Group B; Pazopanib + Pemetrexed - Group C

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of the combination of Xalkori (crizotinib) either with Votrient (pazopanib) or Alimta (pemetrexed) or of the combination of 3 study drugs that can be given to patients with advanced cancer. The safety of these drug combinations will also be studied.

Crizotinib is designed to block a protein called ALK, which is involved in cancer cell growth and survival.

Pazopanib is designed to block the growth of blood vessels that supply nutrients needed for tumor growth. This may prevent or slow the growth of cancer cells.

Pemetrexed is designed to block proteins that may cause tumors to grow.

This is an investigational study. Crizotinib is FDA approved and commercially available for the treatment of locally advanced or metastatic non-small cell lung cancer. Pazopanib is FDA approved and commercially available for treatment of advanced renal cell carcinoma. Pemetrexed is FDA approved and commercially available for the treatment of non-small cell lung cancer.

The combination of crizotinib with pazopanib, crizotinib with pemetrexed, pazopanib with pemetrexed, and giving all 3 drugs together to patients with advanced cancer is investigational.

Up to 364 patients will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Study groups:

Dose escalation:

If you are found to be eligible to take part in this study, your doctor will decide if you will receive one of the following drug combinations:

* If you are in Group A, you will receive crizotinib and pazopanib.
* If you are in Group B, you will receive crizotinib and pemetrexed.
* If you are in Group C, you will receive pazopanib and pemetrexed.
* If you are in Group D, you will receive crizotinib, pazopanib, and pemetrexed.

Once it is decided which combination you will receive, you will be assigned to a dose level based on when you join the study.

Up to 8 dose levels of crizotinib with pazopanib will be tested. Up to 6 dose levels of crizotinib with pemetrexed will be tested. Up to 6 dose levels of pazopanib with pemetrexed will be tested. Up to 8 dose levels of pazopanib with pemetrexed and crizotinib will be tested. Up to 6 participants will be enrolled at each dose level.

The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose combination is found.

Dose expansion:

Once the highest tolerable dose of each study drug combination is found, up to 14 more participants may be enrolled to further study the safety of each combination of drugs at that dose.

Study Drug Administration:

Each study cycle is 21 days. Drugs should be taken and/or administered simultaneously. On days of pharmacokinetic testing (if you agree) you should take the drugs at least 1 hour before or 2 hours after a meal.

If you are taking crizotinib, you will take it by mouth at the same time every day consistently either with or without food. It should be swallowed whole with a glass of water. You will take the drug every other day, 1 or 2 times a day. You will be told how often to take this drug.

If you are taking pazopanib, you will take it by mouth at the same time every day with a glass of water. You should take it at least 1 hour before or 2 hours after a meal.

If you receive pemetrexed:

* You will receive it by vein on Day 1 of each cycle over about 10 minutes.
* The day before your first dose of pemetrexed, you will start taking folic acid to help lower the risk of side effects. Although the study drug is designed to prevent the body from making folic acid that could help cancer grow and spread, some folic acid is needed to prevent side effects in non-cancerous tissue. You will take folic acid by mouth 1 time every day until at least 30 days after you received the last dose of pemetrexed.
* The day before your first dose of pemetrexed, you will receive a vitamin B12 injection. You will receive an injection of Vitamin B12 about every 9 weeks after that. Vitamin B12 is given to help reduce the risks of side effects.
* You will take dexamethasone by mouth 2 times a day on the day before, the day of, and the day after you receive pemetrexed.

Study Visits:

At every study visit, you will be asked about any other drugs or herbal supplements you are taking and about any side effects you may have.

During Cycles 1 and 2, you will have weekly blood (about 1 tablespoon) collected for routine tests.

During Week 1 of Cycles 2 and beyond:

* Your medical history will be recorded, including any cancer symptoms.
* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 1 tablespoon) and urine will be collected for routine tests.
* If your doctor thinks it is needed, you will have an ECG to check your heart function.

Every 6 weeks, or earlier if needed, blood (about 1 tablespoon) will be drawn for tumor marker testing.

After about 6 weeks and then every 2-3 cycles after that, you will have a CT scan, x-ray, MRI scan, and/or PET scan to check the status of the disease. It may be done more often if your study doctor thinks it is needed.

If you are able to become pregnant, you will have a blood (about 1 teaspoon) or urine pregnancy test every 2 cycles or at any time the study doctor thinks it is needed.

Length of Study Participation:

You may continue taking the study drugs for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over once you have completed the end-of-dosing and/or follow-up visits.

End-of-Dosing Visit:

Within 30 days after your last dose of study drugs, you will have an end-of-study visit. If you are having side effects at the time of this visit, you may have follow-up for a longer period of time. At this visit, the following tests or procedures may be performed:

* Your medical history will be recorded, including any cancer symptoms.
* You will be asked if you have had any side effects.
* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 1 tablespoon) and urine will be collected for routine tests.
* Blood (about 1 tablespoon) will be drawn for tumor marker testing.
* If the doctor thinks it is needed, you will have an x-ray, CT scan, MRI scan, and/or PET/CT scan to check the status of the disease.
* If your doctor thinks it is needed, you will have an ECG to check your heart function.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced cancer, either refractory to standard therapy or for which no effective standard therapy that increases survival for at least 3 months is available.
2. Patients must have measurable or evaluable disease, as defined by RECIST 1.1.
3. Women of child-bearing potential and men must agree to use adequate contraception.
4. ECOG performance status of 0 to 2.
5. Adequate organ functions: (Crizotinib plus Pazopanib arm A): Neutrophils > 1000/uL; Platelets ≥ 75,000/uL; Total bilirubin < or= 2 x ULN (upper limit of normal); ALT < or = 2.5 x ULN or < o r= 5 x ULN if liver metastases persist; Serum creatinine < 2 x ULN (Crizotinib plus Pemetrexed arm B, Pazopanib plus Pemetrexed arm C, Crizotinib plus Pazopanib plus Pemetrexed arm D) Neutrophils > 1500/uL; Platelets > or = 100,000/uL; Total bilirubin < or = 2 x ULN (upper limit of normal); ALT < or = 2.5 x ULN or < or = 5 x ULN if liver metastases persist; Calculated GFR > 45 mL/min.
6. Creatinine Clearance: The standard Cockcroft and Gault formula must be used to calculate CrCl for enrollment or dosing. Also include in the pre-treatment or baseline text portion of the protocol, the 'On Study Evaluations or During Treatment' for every Pemetrexed treatment day, and also capture in the study Schedule of Events. No dosage adjustment is needed in patients with creatinine clearance > 45 mL/min. Insufficient numbers of patients have been studied with creatinine clearance <45 mL/min to give a dose recommendation. Therefore, Pemetrexed should not be administered to patients whose creatinine clearance is <45 mL/min.
7. For pemetrexed arms: The ability to interrupt NSAIDs 2 days before (5 days for long-acting NSAIDs), the day of, and 2 days following administration of Pemetrexed.
8. The ability to take folic acid, Vitamin B12, and dexamethasone according to protocol for all pemetrexed arms.
9. Expansion cohort only for arms containing crizotinib: arm A (Crizotinib plus Pazopanib) and arm B (Crizotinib plus Pemetrexed) and arm D (Crizotinib plus Pazopanib Plus Pemetrexed) but not arm C (Pazopanib plus Pemetrexed). Patients must have ALK abnormality including: translocation, ALK amplification, mutation and overexpression as determined by FISH, IHC, qPCR, qRT-PCR, array Comparative Genomic Hybridization or direct sequencing (aCGH). Or patients must have a c-Met abnormality; either c-Met amplification or c-Met mutation or patients must have the ROS1 translocation as determined by FISH.

Exclusion Criteria:

1. Patient receiving any concurrent chemotherapy.
2. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring intravenous antibiotics.
3. Symptomatic congestive heart failure (NYHA Class III or IV), unstable angina pectoris or congenital long QT syndrome.
4. Medical and/or psychiatric problems of sufficient severity to limit full compliance with the study or expose patients to undue risk.
5. Known anaphylactic or severe hypersensitivity to study drugs or their analogs.
6. Patient has failed to recover from any prior surgery within 4 weeks of study entry.
7. Patient is pregnant or lactating.
8. Patient has had any treatment specific for tumor control within 3 weeks of dosing with investigational drugs and cytotoxic agents, or within 2 weeks of cytotoxic agent given weekly, or within 6 weeks of nitrosoureas or mitomycin C, or within 5 half-lives of biological targeted agents with half-lives and pharmacodynamic effects lasting less than 5 days (that includes, but is not limited to, erlotinib, sorafenib, sunitinib, bortezomib, and other similar agents).
9. Patient has any signs of intestinal obstruction.
10. Patient is not able to swallow oral medication.
11. Patients receiving whole brain radiation within 14 days prior to the first dose of study drugs will be excluded. NOTE: Patients receiving palliative radiation (other than whole brain) before or during treatment may still be eligible as long as there are evaluable lesions that are not being irradiated.
12. Pemetrexed arms only: Presence of third space fluid which cannot be controlled by drainage.
13. Additional Exclusions for the 3 pazopanib containing arms (Crizotinib plus Pazopanib) and (Pazopanib plus Pemetrexed) and (Crizotinib plus Pazopanib plus Pemetrexed). 1. History of stroke or transient ischemic attack within 6 months prior to study enrollment. 2. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment. 3. Urine for proteinuria > or = 2+ (patients discovered to have > or = 2+ proteinuria on urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate < or = 1g of protein in 24 hours to be eligible).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-08-26 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Crizotinib and Pazopanib | 4 weeks
  If not more than 33% of participants in cohort develop dose limiting toxicity (DLT), this cohort considered MTD. MTD defined by DLTs that occur in first cycle (4 weeks). DLT defined as: Clinically grade 3 or 4 non-hematologic toxicity. Grade 4 hematologic toxicity lasting 3 weeks or longer. Grade 4 nausea or vomiting > 5 days despite maximum anti-nausea regimens. Grade 3 non-hematologic toxicity including symptoms/signs of vascular leak or cytokine release syndrome; or any severe or life-threatening complication or abnormality not defined in the NCI-CTCAE v4.0 attributable to therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Sarina Piha-Paul, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Subbiah V, McMahon C, Patel S, Zinner R, Silva EG, Elvin JA, Subbiah IM, Ohaji C, Ganeshan DM, Anand D, Levenback CF, Berry J, Brennan T, Chmielecki J, Chalmers ZR, Mayfield J, Miller VA, Stephens PJ, Ross JS, Ali SM. STUMP un"stumped": anti-tumor response to anaplastic lymphoma kinase (ALK) inhibitor based targeted therapy in uterine inflammatory myofibroblastic tumor with myxoid features harboring DCTN1-ALK fusion. J Hematol Oncol. 2015 Jun 11;8:66. doi: 10.1186/s13045-015-0160-2. PMID 26062823
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org